CLINICAL TRIAL: NCT01547819
Title: Imaging the GABAergic System Using 11C-flumazenil PET to Assess the Role of Mild Traumatic Brain Injury in the Development of Post Traumatic Stress Disorder
Brief Title: Mild Traumatic Brain Injury and Post-Traumatic Stress Disorder
Status: Withdrawn | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Other Study IDs: 120082; 12-CC-0082
Record Dates: First submitted 2012-03-06; First posted 2012-03-08 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-12-18

CONDITIONS: Posttraumatic Stress Disorder; Traumatic Brain Injury
Keywords: TBI; Magnetic Resonance Imaging (MRI); PTSD; PET Imaging; 11C-Flumazenil
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Some people who have a traumatic brain injury (TBI) recover completely. Others, however, develop post-traumatic stress disorder (PTSD), with anxiety and depression. Research suggests that levels of a brain chemical called GABA may differ in people with PTSD compared to those without PTSD. Researchers want to see if TBI can affect GABA in the brain and help develop PTSD. To look at the brain, researchers will use imaging studies with the chemical 11C-Flumazenil, which will help the scan show GABA levels in the brain.

Objectives:

- To study the relationship between PTSD and TBI.

Eligibility:

The subjects will be recruited from the Walter Reed National Military Medical Center (WRNMMC).

* Individuals between 18 and 50 years of age who have PTSD and/or had a mild TBI.
* Healthy individuals between 18 and 50 years of age who have no history TBI and no history of PTSD.

Design:

* Participants will be screened with a physical exam and medical history. Urine and breath samples will also be collected.
* Participants will have two imaging studies, on the same day if possible. The first will be a magnetic resonance imaging scan to look at the brain. The second will be a positron emission tomography scan with the study chemical to look at GABA pathways in the brain....

DETAILED DESCRIPTION:
Objective

The primary objective of this study is to investigate the potential role of mild traumatic brain injury (mTBI) in the development of post-traumatic stress disorder (PTSD). We will characterize the central GABAergic system function in patients with PTSD after TBI (TBI-PTSD), subjects with TBI only (TBI-no PTSD), subjects with PTSD only (PTSD-no TBI ), and healthy non-TBI non-PTSD subjects (HC), using PET imaging with (11)C-Flumazenil (FMZ). Our hypothesis is that neuronal and axonal damage due to TBI results in GABAergic system dysfunction which could potentially lead to or contribute to the development of PTSD. We will also correlate the degree of (11)C-FMZ binding abnormalities with time elapsed since the original physical or psychological trauma in TBI-PTSD and PTSD-no TBI patients.

Study Population

Fifty-six male and female adult subjects will be recruited: 14 subjects with PTSD following an episode of non-penetrating mTBI (TBI-PTSD), 14 subjects with mTBI but no history of PTSD (TBI-no PTSD), 14 subjects with PTSD but no history of TBI (PTSD-no TBI), and 14 healthy volunteers (HC) with no PTSD and no history of TBI. The subjects will be recruited from the Walter Reed National Military Medical Center (WRNMMC).

Design

This is a prospective case-control study of the four subject groups mentioned above. Subjects will be stratified according to detailed psychiatric evaluation performed at WRNMMC. Subjects will not be treated with experimental therapies as part of the research study. This study will provide no direct benefit to subjects.

Outcome Measures

The main outcome measure will be (11)C-FMZ binding potential (BP) differences among these four subject groups. Other outcome measures will include Magnetic Resonance Imaging (MRI) anatomical findings and the correlation of (11)C-FMZ binding abnormalities with time elapsed since the original physical trauma in TBI-PTSD group or original psychological trauma in PTSD only group.

ELIGIBILITY:
* All participants must be enrolled in the protocol at Walter Reed National Military Medical Center.

INCLUSION CRITERIA:

TBI-PTSD SUBJECTS:

Subjects in this group must meet the following inclusion criteria:

* Documented diagnosis of non-penetrating mTBI within the last two years.
* Diagnosis of PTSD (which is known to have occurred following the mTBI event) as per the diagnostic criteria followed by protocol number NNMC.2011.0035 at WRNMMC
* Age 18-50 years of age

TBI-no PTSD SUBJECTS:

Subjects in this group must meet the following inclusion criteria:

* No history of PTSD or other major psychiatric disorders
* Mild TBI diagnosis.
* Age 18-50 years of age

PTSD-no TBI subjects:

Subjects in this group must meet the following inclusion criteria:

* No history of TBI
* PTSD diagnosis as per the diagnostic criteria followed by protocol number NNMC.2011.0035 at WRNMMC.
* Age 18-50 years of age

Healthy Control subjects:

Subjects in this group must meet the following inclusion criteria:

* No history of penetrating or non-penetrating head trauma.
* Exclusion of PTSD or other serious psychiatric disorders by psychiatric evaluation as per the diagnostic criteria followed by protocol number NNMC.2011.0035 at WRNMMC
* Age 18-50 years of age

EXCLUSION CRITERIA:

All Subjects:

Subjects are not eligible for participation in this research study if any of the following conditions exist:

* Subjects with history of strokes, brain tumors, seizure and other neurologic problems
* Subjects with serious medical illness such as heart disease, lung disease, kidney disease, a blood disorder like multiple myeloma, diabetes or blood vessel disease.
* Contraindication(s) to MRI scanning, including pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pump, or shrapnel fragments, morbid obesity and severe claustrophobia).
* Pregnant women or women who are breast-feeding.
* History of taking anxiolytics (namely benzodiazepines and barbiturates), anti-depressants or anti-psychotic drugs, unless abstinence for at least 4 weeks prior to the scan.
* History of taking GABAergic drugs such as gabapentin, vigabatrin, tiagabine, lamotrigine, pregabalin and others unless abstinence for at least 4 weeks prior to the scan.
* Blood alcohol concentration >0.0 using a breathalyzer on the day of the scan.
* Evidence of heavy alcohol use based on AUDIT questionnaire (score >8)
* Evidence of drug dependence based on the urine toxicology screen.
* History of previous radiation exposure from any source that, when combined with PET/CT scan, would exceed NIH RSC limits.
* Lifetime or current diagnosis of schizophrenia or other psychotic disorder, or bipolar disorder
* Subjects who cannot give their own consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02-16; Study Completion 2013-12-18

PRIMARY OUTCOMES:
The main outcome measure will be (11)C-FMZ binding potential (BP) in PTSD post mTBI as compared with nTBI without PTSD and healthy control volunteers without PTSD or TBI.

SECONDARY OUTCOMES:
Degree of correlation between 11C-FMZ BP abnormalities and time elapsed since the original physical trauma in TBI-PTSD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Dima A Hammoud, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)

REFERENCES:
- [Background] Rutland-Brown W, Langlois JA, Thomas KE, Xi YL. Incidence of traumatic brain injury in the United States, 2003. J Head Trauma Rehabil. 2006 Nov-Dec;21(6):544-8. doi: 10.1097/00001199-200611000-00009. PMID 17122685
- [Background] Selassie AW, Zaloshnja E, Langlois JA, Miller T, Jones P, Steiner C. Incidence of long-term disability following traumatic brain injury hospitalization, United States, 2003. J Head Trauma Rehabil. 2008 Mar-Apr;23(2):123-31. doi: 10.1097/01.HTR.0000314531.30401.39. PMID 18362766
- [Background] Zaloshnja E, Miller T, Langlois JA, Selassie AW. Prevalence of long-term disability from traumatic brain injury in the civilian population of the United States, 2005. J Head Trauma Rehabil. 2008 Nov-Dec;23(6):394-400. doi: 10.1097/01.HTR.0000341435.52004.ac. PMID 19033832